CLINICAL TRIAL: NCT06564467
Title: A Phase І, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of JMT202 Injection in Chinese Healthy Participants
Brief Title: A Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of JMT202
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JMT202-001
Record Dates: First submitted 2024-07-10; First posted 2024-08-21 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-07

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Intervention Model Description: Drug: JMT202 Other: Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JMT202 SAD experimental group (Experimental): Participants in SAD experimental groups will receive a single subcutaneous injection of JMT202 on Day 1.
  Interventions: Drug: JMT202
- Placebo SAD group (Placebo Comparator): Participants in SAD experimental groups will receive a single subcutaneous injection of placebo on Day 1.
  Interventions: Drug: Placrbo

INTERVENTIONS:
Drug: JMT202 — subcutaneous injection
  Arms: JMT202 SAD experimental group
Drug: Placrbo — subcutaneous injection
  Arms: Placebo SAD group

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single ascending dose (SAD) study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneously Administered JMT202 in Healthy Participants.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 - 60 years (inclusive), male or female;
2. BMI: 18.0-26.0 kg/m^2 (inclusive), with a minimum weight of 50.0 kg (inclusive) for male and 45.0 kg (inclusive) for female;
3. Normal vital signs; Normal physical examination; Normal ECG findings; Normal laboratory examination; Normal imaging examination (X-ray);
4. Participants and their partners agree to use effective and reliable contraceptive methods to avoid pregnancy, and male subjects had no plans to donate sperm, and female subjects had no plans to donate eggs, from the time they signed the informed consent to 6 months after the end of the study;
5. Participants must give informed consent before the trial, fully understand the content, procedures and possible adverse reactions, and voluntarily sign a written informed consent.

Exclusion Criteria:

1. Allergic constitution or known history of allergy to the components of the study drug or similar drugs；
2. Participants with a history of serious diseases, including pancreas, cardiovascular, liver, kidney, blood and lymphatic, central nervous system, and gastrointestinal systems, or other important diseases that may affect the absorption, metabolism, or excretion of the study drug;
3. Participants with a history of cancer, mental illness, depression, anxiety, and epilepsy;
4. With diabetes, thyroid dysfunction or have other affect blood glucose metabolic endocrine disease;
5. HbA1c >6.5% at screening;
6. AST or ALT>1.5 times the upper limit of normal at screening;
7. Fasting triglycerides>1.7 mmol/L at screening;
8. The estimated glomerular filtration rate (eGFR) during screening was < 90 mL/min/1.73 m^2 (calculated by simplified MDRD formula);
9. Screening, vital signs has one or more check exception: temperature < 35.5 ℃ or > 37.2 ℃, pulse < 60 times/min or > 100 times/min, systolic blood pressure ≥ 140 mmHg or < 90 mmHg, diastolic blood pressure ≥ 90 mmHg or < 60 mmHg；
10. During screening, participants with prolonged QT/QTc interval (QTcF > 450 ms in male, > 470 ms in female);
11. Participants with non-negative test for any of HBsAg, HCV antibodies, syphilis antibodies, and HIV antibodies;
12. Blood loss or blood donation of more than 400 mL within 3 months prior to administration;
13. Those who underwent major surgery within 6 months prior to initial administration;
14. Vaccination was administered within 28 days before the trial or within 1 week after the planned dose;
15. Antibody drugs targeting β-Klotho/FGFR1c have been used before screening;
16. Use of any drug for therapeutic purposes within 2 weeks prior to administration or within the 5 half-lives of the drug (whichever is longer), including prescription drugs, over-the-counter drugs or health care products, Chinese herbs;
17. Participated in another study within 3 months before administration; Or plans to participate in another drug trial during the study
18. Those who have any special diet requirements, cannot accept unified diet and schedule；
19. Those who smoked more than 5 cigarettes per day within 3 months prior to screening and/or did not agree to refrain from using any tobacco products during the study;
20. Regular drinkers within 3 months prior to screening, female more than 14 g (i.e.,145 mL wine, 497 mL beer or 44 mL low-alcohol liquor), male more than 28 g (i.e.,290 mL wine, 994 mL beer or 88 mL low-alcohol liquor), or within 48 h before administration taking any alcohol, and/or test positive for breath alcohol；
21. Regular drinkers within 1 months prior to screening, i.e., those who consume excessive amounts of tea, coffee and/or caffeinated beverages (more than 8 cups, 1 cup = 250 mL) per day, and/or do not agree that tea, coffee and/or caffeinated foods, grapefruit and/or grapefruit juice, and/or products containing opium poppy are prohibited during the study;
22. A history of drug abuse, and/or drug use within 3 months prior to screening, and/or positive urine drug screening;
23. There were symptoms such as dermatitis or skin abnormalities in and around the site of administration;
24. Participants who were dizzy with needles, dizzy with blood, unable to tolerate blood collection by venipuncture, or with poor peripheral venous access conditions;
25. Pregnant or lactating women; blood HCG positive, and/or women of childbearing age who have unprotected sex with their partner within 30 days before screening;
26. The researchers think doesn't fit to participate in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
The Number of adverse events (AEs) electrocardiograms | Pre-dose and multiple timepoints no less than 50 days
  To investigate the safety and tolerability by assesment of AEs following administration.
Number of participants with clinically significant change from baseline in vital signs | Pre-dose and multiple timepoints no less than 50 days
Number of participants with clinically significant change from baseline in electrocardiogram (ECG) findings | Pre-dose and multiple timepoints no less than 50 days
Number of participants with clinically significant abnormalities in physical examination | Pre-dose and multiple timepoints no less than 50 days

SECONDARY OUTCOMES:
Area under the concentration-time curve from 0 to the collection time t (AUC0-t) | Pre-dose and multiple timepoints no less than 50 days
Area under the concentration-time curve from 0 to infinity (AUC0-∞) | Pre-dose and multiple timepoints no less than 50 days
Time to maximum concentration (Tmax) | Pre-dose and multiple timepoints no less than 50 days
Serum Maximum concentration (Cmax) | Pre-dose and multiple timepoints no less than 50 days
Half-Life (t1/2) | Pre-dose and multiple timepoints no less than 50 days
Anti-drug antibody (ADA) prevalence in blood before study treatment and at the Follow-up Visit | Pre-dose and multiple timepoints no less than 50 days
Absolute change in High molecular weight adiponectin | Pre-dose and multiple timepoints no less than 50 days
Absolute change in weight | Pre-dose and multiple timepoints no less than 50 days
Absolute change in glycosylated hemoglobin | Pre-dose and multiple timepoints no less than 50 days
Absolute change in fasting insulin level | Pre-dose and multiple timepoints no less than 50 days
Absolute change in fasting glucose | Pre-dose and multiple timepoints no less than 50 days
Absolute change in blood lipoprotein | Pre-dose and multiple timepoints no less than 50 days

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Li, doctor, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijin, China